CLINICAL TRIAL: NCT02860195
Title: Evaluation of the Sensitivity of a Transdermal Device to Monitor the Sweat Alcohol Concentration
Acronym: ALCOOCAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-12; 2016-A00729-42 (Registry Identifier: ANSM)
Record Dates: First submitted 2016-07-27; First posted 2016-08-09 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: The Sweat Alcohol Concentration
MeSH Terms: interventions — Ethanol; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Other: oral dose of alcohol; Device: alcotest; Biological: blood samples; Device: Transdermal monitor

INTERVENTIONS:
Other: oral dose of alcohol
Device: alcotest
Biological: blood samples
Device: Transdermal monitor

SUMMARY:
A non invasive transdermal sensor device was developed by the Im2Np laboratory to determine the presence of vapor of alcohol in insensible perspiration.

One of possible application would be a continuous and non invasive monitoring of drinking behavior. To investigate the validity of this method, it's necessary to compare Transdermal Alcohol Concentrations results obtained by this new device with Blood Alcohol Concentrations and breath Alcohol Concentrations provided by reference methods.

The purpose of this study is to identify the kinetic of alcohol concentration in blood, exhaled air and sweat after alcohol ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-40 years, age-matched (+ 3 years)
* Caucasian
* BMI: 19 to 28 kg/m2
* No smoking or light smoker (<5 cig/d)
* Moderate consumer of alcohol (3-14 drinks/week), with the intoxicated experience

Exclusion Criteria:

* Subjects with addiction to toxic or alcohol (MINI Questionnaire)
* Positive individuals in search of drugs and toxic
* Anxiety or depressive subjects (IASTA Questionnaires and BDI)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The determination of ethanol in the plasma | 6 months
  blood samples

SECONDARY OUTCOMES:
measures in the exhaled air | 6 months
  Assessed with the device Alcotest®
sweat alcohol concentration | 6 months
  assessed with a Transdermal monitor

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille; OLIVIER BLIN, Principal Investigator — ASSISTANCE PUBLQIUE HOPITAUX DE MARSEILLE